CLINICAL TRIAL: NCT01020175
Title: A Phase III, Randomized, Multicentre Trial Comparing Allogeneic Filgrastim Mobilised Peripheral Blood Progenitor Cell Transplantation (PBPCT) With Allogeneic Bone Marrow Transplantation (BMT) in Patients With Acute Leukemia, Chronic Myelogenous Leukemia or Myelodysplastic Syndrome
Brief Title: Peripheral Blood (PB) Versus Bone Marrow (BM) in Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Amgen (Industry); Hoffmann-La Roche (Industry)
Responsible Party: EBMT
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCSF-940136
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Acute Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: allogeneic transplantation; Leukemia; GvHD; MDS
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Leukemia | interventions — Bone Marrow Transplantation; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone marrow transplantation (Other): Patients received bone marrow transplantation
  Interventions: Procedure: Bone marrow transplantation
- Peripheral blood stem cell transplantation (Other): Patients received filgrastim-mobilized peripheral blood stem cell transplantation
  Interventions: Procedure: Peripheral blood stem cell transplantation

INTERVENTIONS:
Procedure: Bone marrow transplantation — Patients received bone marrow transplantation
  Arms: Bone marrow transplantation
Procedure: Peripheral blood stem cell transplantation — Patients received filgrastim-mobilized peripheral blood stem cell transplantation
  Arms: Peripheral blood stem cell transplantation

SUMMARY:
350 patients with early leukemias were assigned to receive peripheral blood or bone marrow transplantation; the occurrence of acute and chronic graft versus host disease, survival, transplantation-related mortality, and relapse rates were compared.

DETAILED DESCRIPTION:
The trial was designed to investigate the safety and outcome of allogeneic filgrastim-mobilized PBPCT compared with allogeneic BMT in patients with standard-risk leukemia. A total of 350 patients between 18 and 55 years of age with acute leukemias in remission or chronic myelogenous leukemia in first chronic phase were randomized to receive either filgrastim-mobilized peripheral blood progenitor cells or bone marrow cells from HLA-identical sibling donors after standard high-dose chemoradiotherapy. The study was approved by the ethics committees of all participating centers, and all patients and donors gave informed consent before any study-related procedure was performed. Donor-recipient pairs were randomized to undergo either BMT or PBPCT. Randomization was carried out centrally at the International Institute for Drug Development (id2), Brussels, Belgium, and used the minimization method to allocate donor and recipient to allogeneic BMT or PBPCT. The randomization strata were as follows: diagnosis (chronic myeloid leukemia [CML] vs other diseases), sex mismatch of donor and recipient, and whether the donor was female and nulliparous. Follow-up visits were scheduled for 6, 12, 24, and 36 months after the date of transplantation.

Neutrophil and platelet recovery occurred significantly faster after transplantation of peripheral blood progenitor cells than after bone marrow transplantation. Acute graft versus host disease of grades II-IV was significantly more frequent in recipients of peripheral blood progenitor cells than in recipients of marrow cells The cumulative incidence of chronic graft versus host disease was higher with peripheral blood progenitor cells than with bone marrow cells

ELIGIBILITY:
Inclusion Criteria:

* Patients with either diagnosis of AML in first or second remission, in first untreated relapse (blast count in marrow < 30%); ALL in first or second remission, in first untreated relapse (blast count in marrow < 30%); CML in first chronic phase, in first accelerated phase (total blast and promyelocytes in marrow and or peripheral blood < 30%) or MDS (excluding RAEB-t).
* Age between 18 and 55 years.
* ECOG performance status between 0,1 or 2.
* HLA-identical sibling donor.
* Written informed consent.

Exclusion Criteria:

* Serum creatinine more than 10% above the normal range for the centre.
* Left ventricular size and function abnormal.
* DLCO < 50%.
* Bilirubin > 2mg/dL (34.2 µmol/L).
* Splenectomised or splenic irradiation.
* Psychiatric, addictive, or any other disorder, which compromises ability to give truly informed consent for participation in this study.
* Currently receiving non-licensed drugs which may affect GVHD or engraftment.
* Pregnant or lactating women.
* Known sensitivity to E.coli derived products.
* HIV positive.
* Previously received BM/PBPC transplant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 1995-01; Primary Completion 1999-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
The primary end point of the study was the maximum grade of acute graft versus host (GVH) disease observed in the recipient.

SECONDARY OUTCOMES:
Incidence of acute GVH disease grade II or above
Time to acute GVH disease
Time to an unsupported platelet count of 20 _ 109/L and 50 _ 109/L
Time to absolute neutrophil count (ANC) of 0.5 x 10e9/L and 1 x 10e9/L
Incidence and severity of chronic GVH disease
Leukemia-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Nobert Schmitz, Prof., Study Chair — Christian-Albrechts- Universita¨t, Kiel, Germany; H Greinix, Dr, Principal Investigator — Allgemeines Krankenhaus, Vienna, Austria; D Niederwieser, Dr, Principal Investigator — University Hospital Innsbruck, Austria; M. Boogaerts, Dr., Principal Investigator — University Hospital, Leuven, Belgium; A Ferrant, Dr, Principal Investigator — Cliniques Universitaires St Luc, Brussels, Belgium; R. Arnold, Dr., Principal Investigator — Charite der Humboldt Universität, Berlin, Germany; E Gluckman, Dr., Principal Investigator — Hopital St Louis, Paris, France; N C Gorin, Dr., Principal Investigator — Hoˆpital St Antoine, Paris, France; N Frickhofen, Dr, Principal Investigator — Universita¨t Ulm, Germany; P Dreger, Dr., Principal Investigator — Christian-Albrechts- Universita¨t, Kiel, Germany; A Zander, Dr, Principal Investigator — Universitätsklinikum Eppendorf, Hamburg, Germany; S McCann, Dr., Principal Investigator — St James Hospital, Dublin, Ireland; A Nagler, Dr., Principal Investigator — Hadassah University Hospital, Jerusalem, Israel; A Bacigalupo, Dr., Principal Investigator — Ospedale San Martino, Genova, Italy; A Gratwohl, Dr., Principal Investigator — Kantonsspital, Basel, Switzerland; J Apperley, Prof., Principal Investigator — Hammersmith Hospital, London, United Kingdom; N H Russell, Dr., Principal Investigator — Nottingham City Hospital, United Kingdom; O Ringde´n, Dr., Principal Investigator — Huddinge Hospital, Sweden; I Majolino, Dr., Principal Investigator — Ospedale V Cervello-USL, Palermo, Italy; J P Jouet, Dr., Principal Investigator — Hopital Claude Huriez, Lille, France; B Varet, Dr., Principal Investigator — Hopital Necker, Paris, France; J Finke, Dr., Principal Investigator — Klinikum der Albert-Ludwigs-Universität, Freiburg, Germany; G. Smith, Dr., Principal Investigator — Leeds General Infirmary, United Kingdom; A Bosi, Dr., Principal Investigator — Azienda Ospedaliera Careggi, Firenze, Italy; G Lambertenghi-Deliliers, Dr., Principal Investigator — Padiglione G Marcora, Ospedale Maggiore di Milano, Italy; K Kolbe, Dr., Principal Investigator — Universitatsklinikum, Mainz, Germany; T Ruutu, Dr., Principal Investigator — Helsinki University CT. Rentral Hospital, Finland; K A Bradstock), Dr., Principal Investigator — Westmead Hospital, Australia; B Lioure, Dr., Principal Investigator — LCHRU de Hautepierre, Strasbourg, France; T Hughes, Dr., Principal Investigator — Hanson Centre for Cancer Research, Royal Adelaide Hospital, Australia; J Szer, Dr., Principal Investigator — Royal Melbourne Hospital, Parkville, Australia; R Herrmann, Dr., Principal Investigator — Royal Perth Hospital, Australia; L Tru¨mper, Dr., Principal Investigator — Universitätsklinik, Homburg, Germany; M Falda, Dr., Principal Investigator — Centro Dipartimentale Trapianti di Midollo, Ospedale Molinette, Torino, Italy; M Beksac, Dr., Principal Investigator — Ankara University Medical Facility, Turkey; E Nikiforakis, Dr., Principal Investigator — Evangelismos General Hospital, Athens, Greece; M Abecasis, Dr., Principal Investigator — Instituto Portugues de Oncologia Francisco Gentil, Lisboa, Portugal; J Rowe, Dr., Principal Investigator — Rambam Medical Center, Haifa, Israel; M Potter, Dr., Principal Investigator — Royal Free Hospital Hampstead, London, United Kingdom; H Wandt, Dr., Principal Investigator — Medizinische Klinik Nurnberg, Germany; R Schwerdtfeger, Dr., Principal Investigator — Stiftung Deutsche Klinik f. Diagnostik, Wiesbaden, Germany; J Casper, Dr, Principal Investigator — University Rostock, Germany; A. Pagliuca, Dr., Principal Investigator — King's College Hospital, London, United Kingdom
Locations (1):
- Dr. Norbert Schmitz, Hamburg, Germany

REFERENCES:
- [Derived] Friedrichs B, Tichelli A, Bacigalupo A, Russell NH, Ruutu T, Shapira MY, Beksac M, Hasenclever D, Socie G, Schmitz N. Long-term outcome and late effects in patients transplanted with mobilised blood or bone marrow: a randomised trial. Lancet Oncol. 2010 Apr;11(4):331-8. doi: 10.1016/S1470-2045(09)70352-3. Epub 2010 Jan 30. PMID 20117965